CLINICAL TRIAL: NCT04655014
Title: Effects of High Intensity Circuit Training on Physical Fitness, Body Fat Percentage and Waist-Hip Ratio Among Sedentary Females of Sikandarabad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Sana Mehmood, Principal Investigator, Ziauddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sana Mehmood
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Circuit Training (Experimental): The High Intensity Circuit Training comprises of 7 full body exercises as per recommendation of ACSM Where the participants shall be given total of 18 sessions of their respective protocol, comprising of 20 minutes, 3 times/ week for duration of six weeks
  Interventions: Other: High Intensity Circuit Training

INTERVENTIONS:
Other: High Intensity Circuit Training — The High Intensity Circuit Training comprises of 7 full body exercises as per recommendation of ACSM Where the participants shall be given total of 18 sessions of their respective protocol, comprising of 20 minutes, 3 times/ week for duration of six weeks

SUMMARY:
Globally, insufficient Physical Activity (PA) and sedentary life style is recognized as major causes of mortality among young and older adults. Approximately, 5 million deaths are attributed due to physical inactivity (PI), which contributes around 6% of global death. The recent evidence shows that 80 million individuals in Pakistan suffered with non-communicable diseases, due to PI that ultimately lead to sedentary behavior. Therefore, the clinical practitioners have been highlighting in improving the physical activity among young adults not only to prevent chronic disease but also to reduce the risk factors. Despite of the fact, a large number of young adults are PI where this proportion remains high among women. WHO reports that generally, PI is found to be more prevalent in women, due to workload of house chores and care giving role in influence of cultural expectations, especially in low socio economic status. Furthermore, several other factors including high cost of fitness programs, access to physical activity facilities, transportation and most importantly time barrier are the major cause of insufficient PA. Addressing the above barriers, different exercise training protocols have been developed to reduce weight in short span of time and then to maintain it. According to American College of Sports Medicine (ACSM), High Intensity Circuit Training (HICT) is a circuit-style workout that uses individual body weight as a resistance therefore eliminating the need of expensive gym equipment such as dumbbells, barbells kettle bells and many more. In addition, HICT can be performed in any environment (at home, parks and in small place) as per the feasibility of the person. However, overweight and obese women are found to adhere easily with short bout of exercises (10 minutes) then same women with long duration of exercises. Therefore, the aim of this study is to provide cost effective and efficient exercise intervention that may not only reduce the disease burden but also motivate young sedentary females for group activity.

DETAILED DESCRIPTION:
A total 60 healthy sedentary overweight females will be recruited from Sikandrabad. The participants shall be screened by using standardize Physical Activity Readiness Questionnaire (PAR-Q & YOU). After screening, a healthy participant will be allowed to attend the orientation session, where a qualified and trained instructor shall discuss and describe the exercise training protocol. The High Intensity Circuit Training comprises of 7 full body exercises as per recommendation of ACSM, where the participants shall be given total of 18 sessions of their respective protocol, comprising of 20 minutes, 3 times/ week for duration of six weeks. Pre and post assessment will be performed for each participant on all three quantitative outcome measures; Physical Fitness, Body fat percentage and Waist-hip ratio. The training protocol will be terminated on the happening of following event; a) Decrease in oxygen saturation < 90%assessed b) Increase in Heart Rate above the highest limits of Targeted Heart Rate c) if subject feel any discomforts, dizziness, fainting or difficulty in breathing during performance.

ELIGIBILITY:
Inclusion Criteria

* Female Participants with a BMI > 25-29 kg/mm2
* Aged 18-35 years.
* Subjects having a sedentary lifestyle, performing only activities of daily living without engaging in any previous exercise training protocol throughout the week, evaluated by Rapid Assessment Disuse Index (RADI) Questionnaire.

Exclusion Criteria

* History of recent surgeries or trauma that hinders in performing high impact exercises.
* Severe orthopedic, musculoskeletal, cardiopulmonary, neurovascular, psychiatric, inflammatory, metabolic, or endocrine diseases and taking any prescribed medications.
* Pregnant females and nursing mothers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage [Pre-treatment] | six weeks
  The body fat composition will be obtained by measuring three-site skin fold thickness including triceps, supra-Ilium and thigh by using the skin fold thickness caliper.
Body Fat Percentage [Post-treatment] | six weeks
  The body fat composition will be obtained by measuring three-site skin fold thickness including triceps, supra-Ilium and thigh by using the skin fold thickness caliper.
Waist-Hip ratio [Pre-treatment] | six weeks
  Waist-hip ratio will be taken with the help of measuring tape by dividing the circumference of waist in centimeters and circumference of hip in centimeters.
Waist-Hip ratio [Post-treatment] | six weeks
  Waist-hip ratio will be taken with the help of measuring tape by dividing the circumference of waist in centimeters and circumference of hip in centimeters.
Physical Fitness [Pre-treatment] | six weeks
  The Modified Harvard step test is used to measure Physical fitness by dividing duration of exercise and pulse count between 1 and 1.5 seconds.
Physical Fitness [Post-treatment] | six weeks
  The Modified Harvard step test is used to measure Physical fitness by dividing duration of exercise and pulse count between 1 and 1.5 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No